CLINICAL TRIAL: NCT00592696
Title: TRIAD Project: Qualitative Study of Adolescent Depression and Smoking
Status: Completed | Type: Observational
Sponsor: Drexel University College of Medicine (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Suzanne Levy, Investigator, Drexel University
Organization: Drexel University (Other)
Other Study IDs: 16039
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Adolescent - Emotional Problem; Smoking
Keywords: Adolescent depression; Adolescent smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation

SUMMARY:
It has been shown in the adult literature that smoking is related to depression and visa versa. Not much is known about how this relationship is started or if one perhaps leads to the other. We are performing 1 hour long interviews with adolescents ages 12-19 who meet criteria for major depression and who smoke. They are interviewed along with their parent. Questions center around their view of depression and their history of depression as well as questions around their smoking as well as the interrelationships between the two. Transcripts are made of the interview and are being analyzed for themes.

ELIGIBILITY:
Inclusion Criteria:

* 12-19 years old
* Major depression
* Smoke cigarettes
* Lives with parents
* No confidentiality issues related to smoking

Exclusion Criteria:

* Non English speaking
* Suicidal ideation
* Pregnant

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents ages 12-19 who live with their parental guardian who meet criteria for major depression and who smoke cigarettes.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-12; Primary Completion 2008-05 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To determine relationships that exist between smoking and depression in adolescents | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Don Schwarz, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- St. Christopher's Hospital for Children, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Levy SA, Westin AM, Reamy AM, Reyner JC, Syed T, Diamond GS. Communication about smoking between depressed adolescents and their parents. Nicotine Tob Res. 2010 Mar;12(3):191-7. doi: 10.1093/ntr/ntp192. Epub 2010 Jan 6. PMID 20053789